CLINICAL TRIAL: NCT00972530
Title: The Importance of Immobilisation After Intra-articular Glucocorticoid Treatment for Elbow Synovitis - a Randomised and Controlled Study
Brief Title: Intra-articular Glucocorticoid Treatment of the Elbow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Gävleborg (Other)
Collaborators: Meda AB (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dnr 2005:362
Record Dates: First submitted 2009-09-03; First posted 2009-09-07 (Estimated); Results first posted 2009-11-11 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2009-10

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; treatment
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Immobilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Activity (No Intervention): Normal activity without restrictions
- immobilisation (Active Comparator): 48 hours postinjection rest
  Interventions: Behavioral: immobilisation in a triangular sling

INTERVENTIONS:
Behavioral: immobilisation in a triangular sling — Intervention group: Immobilisation 48 hours in a triangular sling (mitella)
  Control group: normal activity without restrictions
  Other Names: Postinjection rest; normal joint usage
  Arms: immobilisation

SUMMARY:
BACKGROUND: Intra-articular glucocorticoid injections are frequently used to relieve symptoms of arthritis. Postinjection rest has been shown to improve the outcome of knee joint injections, but not for wrist injections. Consequently, different joints respond differently on postinjection regimens.

OBJECTIVES: To investigate whether better treatment results might be achieved of post-injection rest following intra-articular glucocorticoid treatment for elbow synovitis.

METHODS: 90 patients with rheumatoid arthritis (RA) and elbow synovitis were treated with 20 mg intra-articular triamcinolone hexacetonide and randomised to either a 48 hour immobilisation in a triangular sling (n=46) or normal activity without restrictions (n=44). Primary endpoint was relapse of synovitis. In addition, pain, function according to a self assessment questionnaire (PREE) and range of movement were followed for six months.

ELIGIBILITY:
Inclusion Criteria:

* Rheumatoid arthritis, and
* Clinical signs of elbow synovitis

Exclusion Criteria:

* Patients in function class 4 according to Steinbrocker as well as patients with oral glucocorticoid treatment corresponding to more than 7.5 mg prednisolone or intra-articular treatment in the joint the past three months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Weitoft, MD PhD, Principal Investigator — Department of Research and Development County Council of Gävleborg/Uppsala University

REFERENCES:
- [Derived] Weitoft T, Forsberg C. Importance of immobilization after intraarticular glucocorticoid treatment for elbow synovitis: a randomized controlled study. Arthritis Care Res (Hoboken). 2010 May;62(5):735-7. doi: 10.1002/acr.20039. PMID 20461791

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Activity | Immobilisation
Started | 44 | 46
Completed | 44 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Activity | Immobilisation | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 31 | 28 | 59
  >=65 years | 12 | 18 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (15.2) | 59.0 (14.6) | 59.3 (14.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 6 | 12 | 18
Region of Enrollment [Number; unit: participants]
  Sweden | 44 | 46 | 90

OUTCOME MEASURES:

1. Primary Outcome: Relapse of Arthritis
Description: The patients were followed for six months and if signs and symptoms recurred in between the patients were told to contact the rheumatology department. In such cases the elbow was re-examined and if a relapse could be confirmed the duration of effect was recorded and if needed the patient was offered another injection.
Time Frame: Regular visits at one week, 3 months and 6 months.
Measure: Number; unit: participants
Arm/Group | Activity | Immobilisation
Number analyzed (Participants) | 44 | 46
participants
  Relapse | 8 | 13
  Mobility one week | 44 | 46
  Mobility 3 months | 43 | 43
  Mobility 6 months | 42 | 41
  Pain one week | 44 | 45
  Pain 3 months | 43 | 43
  Pain 6 months | 42 | 41
  Function one week | 44 | 46
  Function 3 months | 43 | 43
  Function 6 months | 42 | 41

ADVERSE EVENTS:
Arm/Group | Activity | Immobilisation
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46
Other Adverse Events (participants affected / at risk) | 0/44 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No